CLINICAL TRIAL: NCT06398106
Title: Proactive Therapeutic Drug Monitoring Versus Routine Care With the Novel Biologics in Psoriasis : a Pragmatic, Multicentric, Randomised, Controlled Study
Brief Title: Proactive TDM Versus Standard Use of Biologics in Psoriasis
Acronym: HELIOS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2024-0151; 2023-509637-39-00 (EU CTIS Number); KCE-22-1375 (Other Grant/Funding Number: KCE)
Record Dates: First submitted 2024-04-24; First posted 2024-05-03 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Psoriasis Vulgaris
Keywords: Therapeutic drug monitoring; Biologics
MeSH Terms: interventions — secukinumab; ixekizumab; guselkumab

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard dosing of biologics (No Intervention): Patients will receive biological therapy according to standard clinical practice. Secukinumab, ixekizumab and guselkumab will be administered according to standard dosing regimen. Adjustments in doses and intervals, or biological switch according to clinical parameters or at the physicians' discretion are considered as standard clinical practice.
  Investigators will not have access to information on levels of the drug or antidrug antibodies and no decision tree will be provided to guide treatment adjustments.
- Proactive TDM based dosing (Experimental): Stepwise treatment modifications based on drug levels: if the drug level is below/above the target the dose of the biologic will be increased/decreased by stepwise interval shortening/lengthening - first modified by 33% and then 50% increase or decrease. If the target is still not reached at the next study visit, the dosing interval will be shortened or prolonged with one additional week at each additional visit until the target is reached.
  In case the dosing regimen shifts from dose increase to dose decrease or vice versa, the dosing interval will be shortened or prolonged with one additional week at each additional visit until the target is reached.
  Interventions: Drug: Proactive TDM-based dosing of secukinumab; Drug: Proactive TDM-based dosing of ixekizumab; Drug: Proactive TDM-based dosing of guselkumab

INTERVENTIONS:
Drug: Proactive TDM-based dosing of secukinumab — Maintenance/normal dose is 300 mg/4 weeks.
  First dose reduction step: 300 mg/6 weeks. Second dose reduction step: 300 mg/8 weeks. Further dose reduction steps: prolongation with 1 additional week
  First dose escalation step: 300 mg/3 weeks Second dose escalation step: 300 mg/2 weeks Further dose escalation step: shortening with 1 additional week
  Other Names: Cosentyx
  Arms: Proactive TDM based dosing
Drug: Proactive TDM-based dosing of ixekizumab — Maintenance/normal dose is 80 mg/4 weeks.
  First dose reduction step: 80 mg/6 weeks. Second dose reduction step: 80 mg/8 weeks Further dose reduction steps: prolongation with 1 additional week
  First dose escalation step: 80 mg/3 weeks Second dose escalation step: 80 mg/2 weeks Further dose escalation step: shortening with 1 additional week
  Other Names: Taltz
  Arms: Proactive TDM based dosing
Drug: Proactive TDM-based dosing of guselkumab — Maintenance/normal dose is 100 mg/8 weeks.
  First dose reduction step: 100 mg/12 weeks. Second dose reduction step: 100 mg/16 weeks. Further dose reduction steps: prolongation with 1 additional week
  First dose escalation step: 100 mg/6 weeks Second dose escalation step: 100 mg/4 weeks Further dose escalation step: shortening with 1 additional week
  Other Names: Tremfya
  Arms: Proactive TDM based dosing

SUMMARY:
Biologics are effective agents for the treatment of psoriasis. The newest generation of biologics block interleukin 17 and 23. Physicians always prescribe these drugs in a fixed dose, but this may lead to under- and overdosing in some patients. Underdosing may lead to inadequate response or loss of response over time. Overdosage, on the other hand, can lead to higher risk of side effects and higher costs for the healthcare system. In daily clinical practice, physicians often tackle this real-world issue by blind trial- and- error dose modifications or switching to another biologic. In this study, we want to rationalize these dose modifications and optimize dosing based on the drug concentrations, measured in the blood of the patient (i.e. therapeutic drug monitoring). Depending on the drug concentration, the interval between injections will be lengthened or shortened with the aim to reach the required drug concentration to reach the best clinical result. The trial will be conducted in 14 Belgian hospitals where patients will be divided into 2 study groups: a group that will be advised on the dosing scheme of their biologic based on the measured drug concentration and a group that continues dosing as in daily clinical practice. We will monitor if the clinical response and quality of life remains stable. With this study, we will track drug concentrations as we believe that they can guide dosing of biologics and we hope to achieve better safety, lower healthcare expenses and higher patients' treatment satisfaction while striving for the best clinical response.

DETAILED DESCRIPTION:
Rationale:

Biologics are effective agents for the treatment of psoriasis. The newest generation of biologics block interleukin 17 and 23. Physicians always prescribe these drugs in a fixed dose, but this may lead to under- and overdosing in some patients. Underdosing may lead to inadequate response or loss of response over time. Overdosage, on the other hand, can lead to higher risk of side effects and higher costs for the healthcare system. In daily clinical practice, physicians often tackle this real-world issue by blind trial- and- error dose modifications or switching to another biologic. In this study, we want to rationalize these dose modifications and optimize dosing based on the drug concentrations, measured in the blood of the patient (i.e. therapeutic drug monitoring).

Objectives: The primary goal is to assess if proactive TDM is non-inferior compared to standard of care with respect to sustained disease control, defined as an absolute PASI ≤ 2 OR a delta PASI from baseline ≥ 50% during at least 80% of all 3-monthly study visits over a period of 18 months, in patients with moderate to severe psoriasis treated with novel biologics (secukinumab, ixekizumab or guselkumab). Secondary goals are:

To compare proactive TDM to standard of care with respect to disease activity, quality of life, treatment satisfaction and costs of treatment (cost-effectiveness) To identify baseline predictors for sustained disease control. To evaluate the cost-effectiveness of proactive TDM To evaluate the safety of proactive TDM.

Study design: A multicentre, pragmatic, randomised, controlled, non-inferiority trial.

Study population:

Patients with moderate-to-severe psoriasis, treated with secukinumab or ixekizumab (IL-17 inhibitors) or guselkumab (IL-23 inhibitor) in daily clinical practice for at least 6 months on standard dosing (maintenance phase). A total of 210 patients will be randomized (1:1) to the intervention group (TDM based dosing) or continuation of usual care.

Intervention: Stepwise treatment modifications based on drug levels: if the drug level is below/above the target, the dose of the biologic will be increased/decreased by stepwise interval shortening/lengthening - first modified by 33% and then 50% increase or decrease. If the target is still not reached at the next study visit, the dosing interval will be shortened or prolonged with one additional week at each additional visit until the target is reached.

In case the dosing regimen shifts from dose increase to dose decrease or vice versa, the dosing interval will be shortened or prolonged with one additional week at each additional visit until the target is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Adults; aged 18 years or older
2. Documented diagnosis of psoriasis (predominantly type vulgaris; based on clinical diagnosis) by an accredited dermatologist
3. Patients must be currently treated with secukinumab, ixekizumab or guselkumab ≥ 6 months according to the standard dosing scheme.
4. The subject signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any study procedures

Exclusion Criteria:

1. Another indication than plaque psoriasis as the main indication for biologic use (e.g. receives biologic for rheumatoid arthritis as the main indication)
2. Concomitant use of systemic immunosuppressants other than methotrexate or acitretin (e.g. prednisone, cyclosporine etc)
3. Severe comorbidities with short life-expectancy (e.g. metastasized tumour) or uncontrolled PsA at inclusion/baseline
4. Presumed inability to follow the study protocol
5. Active pregnancy wish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of sustained disease control | 18 months
  Sustained disease control, defined as an absolute PASI ≤ 2 OR a delta PASI from baseline ≥ 50% during at least 80% of all 3-monthly study visits over a period of 18 months.

SECONDARY OUTCOMES:
Psoriasis disease activity, measured with the Psoriasis Area and Severity Index (PASI) at each 3-monthly study visit. | 18 months
  Change from baseline at 18 months in PASI score. The PASI measures disease activity. The scores ranges from 0 (skin lesion free) to 72 with higher scores indicating higher disease activity.
Dermatology-related quality of life as measured with the Dermatology Life Quality Index (DLQI-R) at each 3-monthly study visit. | 18 months
  Change from baseline at 18 months in DLQI_R score. The DLQI_R measures QoL. The score ranges from 0 (no impact) to 30 (greatest impact) with higher scores indicating higher impact on quality of life.
Health status of participants, assessed by using the Short Form 36 (SF-36) version 2 questionnaire at every 3-monthly time point. | 18 months
  Change from baseline at 18 months in SF-36 score. The SF-36 measures QoL. The score ranges from 0 (maximum disability) to 100 (no disability). In the field of dermatology, the SF36 has been proposed as the instrument of choice for evaluating QoL in a generic way by Both et al.. Although we acknowledge that the SF36 can be perceived as more difficult to fill in by the patients, comparison of QoL measures by Fernandez-Penas et al, showed that SF-36 was more sensitive than other instruments in detecting worse QoL in male patients. The minimal clinical important difference (MCID) for SF-36 is considered 10 units.
Whether participants will have serious adverse events (SAE) and adverse events of special interest (AEoSI) during the study period. | 18 months
  AEoSI include, but are not limited to,
  * occurrence of infusion reactions
  * drug (biologic) Immunogenicity
  * Moderate-to severe infections
  * Newly diagnosis of cancer
  * New-onset of psoriatic arthritis
  * joint complains
Pharmacokinetics of the drugs of interest | 18 months
  Drug concentrations of each included drug, measured in blood serum samples which will be collected from participants at each 3-monthly time point.
  The drug concentrations will be evaluated with an enzyme-linked immunosorbent assay (ELISA) and compared to the target/reference concentration. In the intervention group, these drug concentrations will guide the modification of the dosing interval (according to a predefined decision tree).
Immunogenicity of the drugs of interest | 18 months
  Anti-drug antibody levels of each included drug, measured in blood serum samples which will be collected from participants at each 3-monthly time point.
Utilities, derived from EuroQoL 5 Dimensions (EQ-5D-5L) questionnaires, which will be measured at each 3-monthly time point. | 18 months
  Utility scores will be used to calculate quality adjusted life years (QALYs) which are used to determine cost-effectiveness of the intervention.
Volumes of care, as measured with the iMTA Medical Consumption Questionnaire (MCQ) at each 3-monthly time point. | 18 months
  The iMTA Medical Consumption Questionnaire (iMCQ) is an instrument for measuring medical consumption. The iMCQ includes questions related to frequently occurring contacts with health care providers. The iMCQ is a generic questionnaire and will be used to calculate direct medicals costs and non-medical costs.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, Prof., Principal Investigator — University Hospital, Ghent
Locations (13):
- Belgium (13):
  - AZ Sint-Jan, Bruges
  - UCL Saint-Luc, Brussels
  - ULB Erasme, Brussels
  - UZ Brussel, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - AZ Alma, Eeklo
  - Dermatologiepraktijk huidziekten Geel, Geel
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - Clinique André Renard, Herstal
  - Dermatologie Handelskaai, Kortrijk
  - UZ Leuven, Leuven
  - Dermatologie Maldegem, Maldegem

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the PsoGent research group — https://psogent.ugent.be/projects.html